CLINICAL TRIAL: NCT00005244
Title: Anger Expression, Self-focus and Coronary Heart Disease Risk Factors
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1125; R01HL041865 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To identify behavioral factors underlying the development of cardiovascular risk in young adults.

DETAILED DESCRIPTION:
BACKGROUND:

The continued number of observations relating the Type A behavior pattern to coronary heart disease underscores the importance of developing a careful theoretical basis that may account for the virulent components of a coronary-prone personality.

CARDIA or Coronary Heart Disease Risk Development in Young Adults is a prospective, epidemiological study of coronary heart disease risk factors in cohorts of Black and white men and women, 18 to 30 years of age.

DESIGN NARRATIVE:

From each of the baseline tape-recorded Type A/B structured interviews administered in CARDIA, eighteen questions were scored for self-references, perceived pressure, anger experience, and anger expression. The anger measures were related to other measures of anger-in and hostility in order to establish their validity. The interrelationships of these factors were assessed separately for each of the socioeconomic status (SES) categories. A major focus of the analyses was to describe SES differences in how pressure was perceived and how anger was experienced and expressed. The study also assessed how these factors were related to data already collected on psychosocial risk factors and primary risk factors including blood pressure, serum cholesterol, and cigarette smoking.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1989-04; Study Completion 1991-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Scherwitz — University of California at San Francisco